CLINICAL TRIAL: NCT00458770
Title: Study of Hypothalamic Metabolism in Spontaneous Cluster Headache Attacks
Status: Terminated | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique Hopitaux De Marseille (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 2006/22; 2009-A00149-48
Record Dates: First submitted 2007-04-10; First posted 2007-04-11 (Estimated); Last update posted 2014-02-25 (Estimated); Status verified 2014-02

CONDITIONS: Cluster Headache
Keywords: Comparison of a spontaneous acute cluster headache attack and rest (no pain) in ten patients with cluster headache defined with IHS criteria
MeSH Terms: conditions — Cluster Headache

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: position emission transaxial tomography — cerebral position emission transaxial tomography using 18Fluorodeoxyglucose

SUMMARY:
Cluster headache is characterized by unilateral excruciating head pain and autonomic dysfunction. Hypothalamic overactivity was observed in nitrate-induced cluster-headache and in only one case of spontaneous cluster headache 'Sprenger et al, 2004). This prompted the application of hypothalamic deep brain stimulation. The aim of this data is to precise the localisation of the hypothalamic activation.

ELIGIBILITY:
Inclusion Criteria:

* cluster headache in crisis
* no serious illnesses in progress as cancer, autoimmune disease, liver disease
* patient without chronic psychiatric disease excluding moderate and reactional depression
* no demential disease
* no anxious or depressive disease
* no contraindication to PET scan (pregnancy and breast-feeding)
* social security cover
* written informed consent

Exclusion Criteria:

* No effective contraception taken
* unable to realize a decubitus of 15 minutes long

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2009-05; Primary Completion 2011-05 (Actual); Study Completion 2011-05 (Actual)

PRIMARY OUTCOMES:
To confirm the existence of a hypothalamic promoter at the origin of Spontaneous Cluster Headache Attacks | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Anne DONNET, PH, Principal Investigator — Pôle de Neurosciences Cliniques CHU Timone, 204 rue St Pierre, Marseille 13385 cedex 5 France
Locations (1):
- Pôle de Neurosciences Cliniques CHU Timone, Marseille, France